CLINICAL TRIAL: NCT00279539
Title: phVEGF165 GENE TRANSFER TO PROMOTE ANGIOGENESIS IN PATIENTS WITH ISCHEMIC HEART FAILURE
Brief Title: Stem Cell Mobilization and VEGF Gene Transfer for Heart Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never started.
Sponsor: Losordo, Douglas, M.D. (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BB-IND 10442
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2009-06

CONDITIONS: Ischemic Congestive Heart Failure (CHF)
Keywords: Cardiovascular; Gene Therapy; DNA; Stem Cells; Congestive Heart Failure; Coronary Artery Disease; CHF; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Cardiomyopathies | interventions — Vascular Endothelial Growth Factor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Vascular Endothelial Growth Factor (VEGF1)

SUMMARY:
The purpose of this study is to evaluate the safety and bioactivity of intramyocardial gene transfer using VEGF (vascular endothelial growth factor) in patients with ischemic heart failure. The research treatment of this CHF study will involve the use of an intramuscular injection with a catheter inserted in through the groin to transfer a type of DNA (phVEGF165 gene) to the wall of the heart. Genes (which are part of the DNA molecules) carry instructions to allow the cells to produce specific proteins. Gene transfer or treatment with DNA (a necessary part of all cells) is being studied for the treatment of patients with heart failure. This research therapy, which is experimental and not proven, is designed to try to grow new blood vessels to improve blood flow to areas of the heart that are not receiving enough blood.

DNA is present in all cells and provides the instructions for making proteins. After delivering a piece of DNA containing the vascular endothelial growth factor 1 (VEGF-1) gene (the product being studied) into cells, the cells may produce a specific protein called vascular endothelial growth factor 1 (VEGF-1). Animal studies have indicated that the VEGF-1 protein may cause new blood vessels to grow. The Vascular Endothelial Growth Factor Gene (ph VEGF 165) is found on the VEGF DNA. Experiments performed in animals show that once in the heart wall, the DNA directs the cells of the heart muscle to make the VEGF protein. VEGF 165 is a protein that has been shown to stimulate cells (known as endothelial cells), which form the inner lining of blood vessels. This protein causes cells to divide and grow, thereby forming new blood vessels. It is anticipated that this new blood supply may help the heart pump the blood more effectively and relieve some heart failure symptoms. We do not yet have enough information to know what will happen in humans, that is why we are doing this research.

After gene transfer we will begin a process to help move some of the stem cells from the bone marrow into the blood circulation. Subjects will be given the drug called G-CSF (a drug used to move cells from the bone marrow into the blood stream). Stem cells are young cells produced by bone marrow (the spongy cavity in the center of large bones) that can develop into blood cells or other types of cells. This medication triggers the movement of stem cells out of the bone marrow and into the blood stream. Before being released into the blood stream, stem cells receive signals that direct them to become specific types of cells such as CD34+ cells (endothelial progenitor cells). CD34+ cells that move to or are in the area of damaged heart tissue may promote growth of new blood vessels that supply blood and nutrients and thereby improve the chance of survival of heart tissue, improve heart function, and possibly have a long-term benefit.

We will be recruiting 12 subjects for this study. There will be no randomization and no placebo group. Once eligibility in the research study has been determined all subjects will be treated with the VEGF and G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Be > 21 years old.
* Have mild or moderate (NYHA Class II or III) CHF secondary to ischemic heart disease.
* Have left ventricular ejection fraction <40%.
* Patients must have total occlusion of one or more extramural coronary arteries demonstrated by diagnostic angiography within 6 months prior to study enrollment.
* Patients must be on a stable cardiac medical regimen (i.e. the same anti-anginal and anti-congestive medications) for 1 month prior to determination of their baseline functional status. The judgment regarding the optimal medical regimen for each individual subject will have been made by the referring cardiologist.
* Subjects must be identified as non-candidates for conventional revascularization by their referring cardiologist.
* Have serum B-type Natriuretic Peptide (BNP) level >100 pg/ml.
* Women of childbearing potential must agree not to become pregnant during the course of the study. Nonsterile men participating in the study must also agree not to impregnate their partners.
* Have the ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

* Have a history of alcohol or drug abuse within 3 months of screening.
* Subjects with evidence (clinical, laboratory, or imaging) or history of neoplasm, or, cancer recurrence within the past 5 years (other than non-melanoma skin cancer or in situ cervical carcinoma).
* Have evidence of moderate to severe proliferative retinopathy on fundoscopic examination by an ophthalmologist.
* History of severe aortic stenosis (aortic valve area < 1.0 cm2) or insufficiency(>2+); severe mitral stenosis (mitral valve area <1.5 cm2); or severe mitral insufficiency(>2+).
* Coronary revascularization procedures within 6 months of study enrollment.
* Documented stroke or transient ischemic attack (TIA) within 60 days of study enrollment.
* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year, such as chronic medical illness (i.e. severe chronic obstructive pulmonary disease, renal failure or cancer).
* Joint or peripheral vascular disease that severely limit treadmill walking.
* Chronic obstructive pulmonary disease that severely limits walking or FEV1.0<30% predicted.
* Have idiopathic or non-ischemic heart failure.
* Have NYHA Class IV heart failure.
* Have or require mechanical ventricular support
* Had surgical heart failure treatments, including left ventricular reconstructive surgery (Dor procedure, cardiomyoplasty, LV banding, etc.)
* Implantation of biventricular pacemaker within 90 days of study treatment.
* Be pregnant or lactating.
* Have a history of an allergy to penicillin.
* Have sickle cell disease.
* Have an untreatable coagulopathy.
* Have a serum creatinine >3.5 mg/dL.
* Have any clinically significant abnormality in liver function or other clinical chemistry or hematology test (defined as a value more than 2 times the upper limit of the normal range for that value).
* Previous enrollment in the study.
* Be unsuitable for participation in the study, in the opinion of the Investigator.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07

PRIMARY OUTCOMES:
LVEF | 6 months
  Left ventricular ejection fraction measured by echo

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Douglas W. Losordo, M.D., Principal Investigator — Northwestern University